CLINICAL TRIAL: NCT03597425
Title: Prognostic Indicators of Survival Following Cardiopulmonary Resuscitation in Patients With Cardiac Arrest: a Single-institutional Study
Brief Title: Prognostic Indicators of Survival Following Cardiopulmonary Resuscitation in Patients With Cardiac Arrest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, GengLong Liu, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: cardiopulmonary resuscitation
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Cardiac arrest; Cardiopulmonary resuscitation; Survival; Prediction
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiopulmonary resuscitation — Cardiopulmonary resuscitation (CPR) is an emergency treatment for patients with respiratory arrest and cardiac arrest in an attempt to restore the patient to spontaneous breathing and heartbeat through cardiopulmonary resuscitation

SUMMARY:
Cardiopulmonary resuscitation (CPR) occurs approximately 200,000 times/yr in hospitals in the UnitedStates, with 18% of patients surviving to discharge. Just over half of these survivors are neurologically intact or with mild defiits at the time of discharge. Do-not-resuscitate (DNR) orders are used to withhold CPR from patients who are unlikely to benefi or for whom it is inconsistent with their treatment goals or personal preferences. It would be helpful to identify patients with a very low likelihood of survival to discharge neurologically intact or with mild defiits were they to experience cardiopulmonary arrest (CPA), so their physician can present the option of a DNR order. This information would also be useful anytime a patient raises the question of the likelihood of survival should they undergo CPA.The objective of this study was to determine key indicators for good outcome in patients with sudden cardiac arrest undergoing CPR and develop a prediction model to predict survival to hospital discharge in these patients.

DETAILED DESCRIPTION:
A CPR coordinator prospectively collected data for the CPR registry according to the Utstein-style guidelines. Te registry included the following information:

demographic data, comorbidities, whether the arrest was witnessed, the incidence of suspected or confrmed trauma, presumed arrest time; presence of bystander CPR, frst documented arrest rhythm by the emergency medical service (EMS) provider, any return of spontaneous circulation (ROSC), presence of ECPR, the presence of return of spontaneous heart beating (ROSB) after CPR, presumed cause of arrest; the application of therapeutic hypothermia and the use of coronary angiography(CAG) or percutaneous coronary intervention (PCI),24-hour survival, the presence of ROSC more than 20 min, hospital length of stay (LOS), survival to hospital discharge,Glasgow-Pittsburgh cerebral performance category (CPC) score at discharge, and the fnal diagnosis at discharge. Te comorbidity score was calculated using the Charlson comorbidity index. Te duration of CPR was defned as the time interval from the frst chest compression provided by healthcare providers to the termination of resuscitation eforts due to ROSC (more than 20 min),ROSB after CPR, or a declaration of death. A favorable neurologic outcome was defned as a CPC score of 1 or 2 on the fve-category scale.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years,
* sudden arrest with potentially reversible causes,
* a short no fow time (time interval from presumed arrest to CPR initiation)
* even for unwitnessed arrests

Exclusion Criteria:

* presence of a terminal illness or malignancy, severe irreversible neurologic defcit,
* suspected or confrmed traumatic origin of arrest,
* no informed consent from the family

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with cardiac arrest
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
indicators of survival | an average of 1 year
  The survival outcome was analyzed with logstic regression

CONTACTS AND LOCATIONS:
Overall Officials: Genglong Liu, Study Chair — Southern Medical University, China
Locations (1):
- Genglong Liu, Shunde, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided